CLINICAL TRIAL: NCT05979298
Title: Open Label Randomized Clinical Study of Plasmid Encoding p62/SQSTM1 (ELenagen) in in Combination With Gemcitabine in Patients With Platinum-resistant Ovarian Cancer
Brief Title: Efficacy of Plasmid Elenagen in Combination With Gemcitabine in Patients With Platinum-resistant Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CureLab Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROC0319
Record Dates: First submitted 2023-07-19; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer; Platinum-resistant Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: This was a prospective randomized multi-center study with two arms. Gemcitabine 1000 mg/m2 days 1,8 every 3 weeks) was administered in both arms: In the Chemo arm (n = 20) GEM was the only treatment, and in the ELENAGEN arm (n = 20) GEM was supplemented with ELENAGEN (2.5 mg i.m. weekly).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabin (Active Comparator): Gemcitabine 1000 mg/m2 days 1,8 every 3 weeks
  Interventions: Drug: Gemcitabine
- Gemcitabine+Elenagen (Experimental): GEM was supplemented with ELENAGEN (2.5 mg i.m. weekly)
  Interventions: Drug: Gemcitabine; Biological: ELENAGEN

INTERVENTIONS:
Drug: Gemcitabine — Chemotherapeutics
  Other Names: Gemzar
Biological: ELENAGEN — DNA plasmid
  Arms: Gemcitabine+Elenagen

SUMMARY:
Phase II, two arm prospective study of efficacy and safety of ELENAGEN in combination with gemcitabine in comparison with gemcitabine alone in patients with platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate safety and efficacy of ELENAGEN, a novel anticancer therapeutics (plasmid DNA encoding p62/SQSTM1) protein, as an adjuvant to chemotherapy with Gemcitabin (GEM) in patients with advanced platinum-resistant ovarian cancer.

This is a prospective randomized multi-center study with two arms. Gemcitabine 1000 mg/m2 days 1,8 every 3 weeks) is administered in both arms: In the Chemo arm (n = 20) Gemcitabine is the only treatment, and in the ELENAGEN arm (n = 20) GEM was supplemented with ELENAGEN (2.5 mg i.m. weekly). The primary endpoint is progression-free survival (PFS), and the secondary endpoint is safety.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18-70 years old.
* Written informed consent of the patient to participate in clinical trials.
* Presence of histologically confirmed ovarian cancer.
* The return of the disease occurred less than 6 months after the last administration of platinum.
* Presence of measurable tumor lesions according to RECIST 1.1 criteria.
* Functional status according to ECOG scale is 0-2.
* Life expectancy of at least 6 months.
* Adequate function of the organs as determined by the following criteria:

  1. Absolute number of neutrophils (ANN) ≥1500/mm3 (≥1.5 × 109/l);
  2. Platelet count ≥100,000/mm3 (IU: ≥100 × 109/l).
  3. Hemoglobin level ≥ 9.0 g/dL determined by analysis performed at least 2 weeks after the last hemotransfusion;
  4. The level of AST and ALT in blood serum not exceeding more than 3 times the upper limit of the norm.
  5. The level of serum bilirubin not exceeding more than 1.5 times the upper limit of normal.
  6. Serum Creatinine ≤ 1.5 mg/dL.
* The ability of the patient to follow the directions of the research physician and follow the study regimen.

Exclusion Criteria:

Criteria by which patients are not included in the study

* Platinum-sensitive relapse of ovarian cancer (disease recurrence occurred more than 6 months after the last administration of platinum drugs).
* Presence of serious diseases or health conditions:

  1. Other malignancies, with the exception of malignancies treated more than 5 years ago without signs of return of the disease.
  2. Brain metastases or leptomeningeal metastases.
  3. Active infection (e.g. fever ≥38 °C), including active or unresolved pneumonia/pneumonitis.
  4. Uncontrolled diabetes mellitus.
  5. Myocardial Infarction in the last 12 months, severe/unstable angina, clinically manifested heart failure class III-IV according to the classification of the New York Cardiology Association (NYCA).
  6. Gastrointestinal bleeding within the last 2 weeks.
  7. Human immunodeficiency virus (HIV), chronic or acute hepatitis B or hepatitis C.
  8. Patients with autoimmune disorders or organ transplantation who require immunosuppressive therapy.

I. Mental illness that may increase the risk associated with participation in the study or taking the study drug or that may affect the interpretation of the results of the study.

K. Polyallergy, bronchial asthma (including aspirin) in history.

* Major surgery during the previous 4 weeks (complete wound healing).
* Previous chemotherapeutic treatment of the patient according to the scheme GEMCITABINE
* Radiotherapy with extended field radiation within the previous 4 weeks or radiotherapy with a limited field radiation within the previous 2 weeks.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer
Enrollment: 40 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years since the start of treatment
  Median duration of time from start of treatment to time of progression by RESIST 1.1 criterion or death

SECONDARY OUTCOMES:
Safety of Elenagen in combination with Gemcitabine | 1 year after the start of treatment
  Frequency of drug-related adverse events (AEs) and serious AEs (SAEs) according to NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Minsk City Clinical Oncology Center, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No
Not to be shared

REFERENCES:
- [Derived] Krasny S, Baranau Y, Bakin E, Polyakov S, Streltsova O, Zharkova E, Filimonava A, Levin G, Gabai V, Shneider A. Elenagen, a p62/SQSTM1-encoding plasmid, improves overall survival in patients with platinum-resistant ovarian cancer: a phase II trial. Int J Gynecol Cancer. 2026 Jan 7:104456. doi: 10.1016/j.ijgc.2025.104456. Online ahead of print. PMID 41577503
- [Derived] Krasny S, Baranau Y, Polyakov S, Zharkova E, Streltsova O, Filimonava A, Siarheyeva V, Kazlouskaya S, Khorau A, Gabai V, Shneider A. Clinical efficacy of plasmid encoding p62/SQSTM1 (Elenagen) in combination with gemcitabine in patients with platinum-resistant ovarian cancer: a randomized controlled trial. Front Oncol. 2024 Feb 12;14:1343023. doi: 10.3389/fonc.2024.1343023. eCollection 2024. PMID 38410116